CLINICAL TRIAL: NCT01181947
Title: VALIANT CAPTIVIA Post-market Registry A Multi-center, Post-market, Non Interventional, Prospective Study
Brief Title: VALIANT CAPTIVIA Post-market Registry
Acronym: VCOUS
Status: Terminated | Type: Observational
Why Stopped: CIP was amended to include long-term FU but, not all sites accepted it so the nr. of pts participating in the extended FU will be small.
Sponsor: Medtronic Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: MDTEV20112009
Record Dates: First submitted 2010-08-10; First posted 2010-08-13 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2023-01

CONDITIONS: Aortic Aneurysm, Thoracic
Keywords: Stent graft; thoracic aorta; dissection; aneurysm; TEVAR; VALIANT; CAPTIVIA; endovascular
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Aneurysm | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients undergoing TEVAR: Those with a thoracic aortic aneurysm/dissection
  Interventions: Device: TEVAR

INTERVENTIONS:
Device: TEVAR — Thoracic endovascular aneurysm repair
  Other Names: Valiant Captivia stent graft system

SUMMARY:
The Valiant Thoracic Stent Graft has been preloaded on the new Captivia Delivery System (Captivia). This new delivery system was CE marked on September 14th, 2009 and was commercially released in the European Union on October 1st, 2009.

The Valiant Thoracic Stent Graft with the Captivia Delivery System (Valiant Captivia) is designed to treat diseases of the descending thoracic aorta including but not limited to aneurysms and dissections.

The purpose of the VALIANT CAPTIVIA Registry is to collect and evaluate mid term clinical performance data of the Valiant Captivia Thoracic Stent Graft System following OUS market approval.

DETAILED DESCRIPTION:
1. Use of controls

   1. This study is a post-market registry without using a control. All analyses will be descriptive in nature and no statistical comparisons are planned.

      Sample size
   2. There is no sample size calculation since this is not a hypothesis driven study; VALIANT CAPTIVIA has recruited 100 subjects and will follow these subjects through for approximately 36 months.
2. Number of investigation sites and study duration

   1. 15 investigation sites in Europe and Turkey where the Valiant Captivia Thoracic Stent Graft System is commercially available have enrolled 100 subjects.
   2. There will be no minimum nor maximum number of enrolled subjects per investigation site.
   3. The sites' compliance with the clinical investigation plan will be assessed on an ongoing basis. In case of serious non-compliance, the sponsor may decide to stop subject enrolment in a site based on the assessment.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years or minimum age as required by local regulations
* Indication for surgical repair of thoracic aortic aneurysms and/or thoracic aortic dissections with an thoracic endovascular stent graft in accordance with the applicable guidelines on endovascular interventions and the Instructions for Use of the Valiant Captivia Thoracic Stent Graft System
* Signed consent form ('Patient informed consent form' or 'Patient Data Release Authorization Form')
* Intention to implant the Valiant Captivia Thoracic Stent Graft System or having implanted the system within the last 3 months before subject enrollment
* Willingness and ability to comply with the CIP

Exclusion criteria

* High probability of non-adherence to physician's follow-up requirements
* Participation in concurrent interventional trial which may confound study results
* Prior implantation of a thoracic stent graft

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Valiant Thoracic Stent Graft with the Captivia Delivery System is indicated for treatment of diseases of the descending thoracic aorta including but not limited to aneurysms and dissections. The Valiant Thoracic Stent Graft is indicated for exclusion of the aneurysm, the false lumen or site of rupture and restoration of blood flow through the stent graft lumen. The device is intended for use in subjects who are candidates for conventional surgical repair, and in subjects who are not candidates for conventional surgical repair due to pre-existing risk factors.
  Study enrolment is open to subjects who in the opinion of the investigator are candidates for endovascular TAA repair with the Valiant Captivia Thoracic Stent Graft System according to the instructions for use (IFU).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Torsello, Prof., Principal Investigator — St Franziskus Hospital GmbH; Rosella Fattori, Prof., Principal Investigator — Policlinico S.Orsola Malpighi; Carlos Vaquero Puerta, Dr., Principal Investigator — Hospital Clínico Universitario de Valladolid; Matthew Thompson, Prof., Principal Investigator — St. George's Hospital; Werner Jaschke, Prof., Principal Investigator — Medical University of Innsbruck; Yigit Goktay, Prof., Principal Investigator — Dokuz Eylul University; Karl Heinz Orend, Prof., Principal Investigator — Universitatsklinikum Ulm; Omke Teebken, Prof., Principal Investigator — Hannover Medical School; Thomas Schmitz-Rixen, Prof., Principal Investigator — Klinikum der J.W.Goethe-Universitat; Markus Steinbauer, Dr., Principal Investigator — Krankenhaus Barmherzige Bruder Regensburg; Stephan Zangos, Dr., Principal Investigator — Klinikum der Johann-Wolfgang-Goethe - Institut fur Diagnostische und Interventionelle Radiologie; Joep Teijink, Dr., Principal Investigator — Catharina Ziekenhuis; Robin Heijmen, Dr., Principal Investigator — St. Antonius Hospital; Mustafa Parildar, Prof., Principal Investigator — Ege University Hospital; Fatih Boyvat, Prof., Principal Investigator — Baskent University Ankara Hospital
Locations (15):
- Medical University of Innsbruck, Innsbruck, Austria
- Germany (6):
  - Klinikum der J.W.Goethe-Universitat, Frankfurt am Main
  - Klinikum der Johann-Wolfgang-Goethe - Institut fur Diagnostische und Interventionelle Radiologie, Frankfurt am Main
  - Medizinische Hochschule Hannover, Hanover
  - St Franziskus Hospital GmbH, Münster
  - Krankenhaus Barmherzige Bruder Regensburg, Regensburg
  - Universitatsklinikum Ulm, Ulm
- Polyclinic Hospital S.Orsola - Malpighi, Bologna, Italy
- Netherlands (2):
  - Catharina Ziekenhuis, Eindhoven
  - St. Antonius Ziekenhuis, Nieuwegein
- Hospital Clinico Universitario de Valladolid, Valladolid, Spain
- Turkey (Türkiye) (3):
  - Baskent University Ankara Hospital, Ankara
  - Dokuz Eylul University, Izmir
  - Ege University Hospital, Izmir
- St George's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Heijmen RH, Thompson MM, Fattori R, Goktay Y, Teebken OE, Orend KH. Valiant thoracic stent-graft deployed with the new captivia delivery system: procedural and 30-day results of the Valiant Captivia registry. J Endovasc Ther. 2012 Apr;19(2):213-25. doi: 10.1583/11-3652MR.1. PMID 22545887

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Undergoing TEVAR: Those with a thoracic aortic aneurysm/dissection>
  > TEVAR: Thoracic endovascular aneurysm repair
Period: Overall Study
Arm/Group | Patients Undergoing TEVAR
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing TEVAR
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 48
Age, Continuous [Median (Full Range); unit: year] | 65.0 [25 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 81
Region of Enrollment [Number; unit: participants]
  Spain | 5
  Turkey | 15
  Austria | 2
  Netherlands | 16
  Germany | 24
  United Kingdom | 21
  Italy | 17
Native aorta diameter [Median (Full Range); unit: mm] | 32 [22 to 42]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success
Description: technical success and freedom from
  * TAA diameter increase of stented segment (>5mm compared to 1 mo),
  * Types I/III endoleak,
  * Aneurysm rupture,
  * Conversion to open surgery,
  * Stent graft occlusion,
  * Stent graft migration resulting in SAE or secondary intervention.
Time Frame: at 12 months
Population: The number of participants analyzed are different for each endpoint based on number of evaluable subjects at each timepoint per endpoint.
Measure: Count of Participants; unit: Participants
Groups:
- 1 - Medtronic VCOUS: TAA Diameter > 5mm at 12 months
- 2 - Medtronic VCOUS: Type I/III Endoleak at 12 months
- 3 - Medtronic VCOUS: Aneurysm Rupture within 12 months
- 4 - Medtronic VCOUS: Stent Graft Occlusion within 12 months
- 5 - Medtronic VCOUS: Conversion to Surgery within 12 months
- 6 - Medtronic VCOUS: Stent Graft Migration > 10 mm resulting in SAE or requiring secondary intervention at 12 months
Arm/Group | 1 - Medtronic VCOUS | 2 - Medtronic VCOUS | 3 - Medtronic VCOUS | 4 - Medtronic VCOUS | 5 - Medtronic VCOUS | 6 - Medtronic VCOUS
Number analyzed (Participants) | 57 | 61 | 100 | 98 | 100 | 64
Participants | 9 | 4 | 4 | 0 | 2 | 1

2. Primary Outcome: Technical Success at Time of Initial Implant
Description: Technical success is defined as successful delivery and deployment of the stent graft (assessed intraoperatively). This is achieved by deployment of the Valiant Thoracic Stent Graft in the planned location with no unintentional coverage of the left subclavian artery, left common carotid artery and/or brachiocephalic artery and with the removal of the delivery system
Time Frame: intraoperatively
Population: The primary and secondary endpoints will be reported descriptively.
  By-gender and by-race data summaries for the primary endpoints, if appropriate, will be generated. Data from all study sites will be grouped together for analyses.
Measure: Number (95% Confidence Interval); unit: participants
Groups:
- Patients Undergoing TEVAR: Those with a thoracic aortic aneurysm/dissection >
  > TEVAR: Thoracic endovascular aneurysm repair
Arm/Group | Patients Undergoing TEVAR
Number analyzed (Participants) | 100
participants | 100 [96.4 to 100.4]

3. Secondary Outcome: SAE
Description: Serious Adverse Events (SAE)
Time Frame: through 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Patients Undergoing TEVAR
Number analyzed (Participants) | 100
participants | 48 [40 to 58]

4. Secondary Outcome: ACM and ARM
Description: All-cause (ACM), Aneurysm related (ARM) and dissection related mortality
Time Frame: at 30 days, 12 months, 24 months and 36 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- 1. VCOUS: Medtronic VCOUS
Arm/Group | 1. VCOUS
Serious Adverse Events (participants affected / at risk) | 48/100
Other Adverse Events (participants affected / at risk) | 5/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. VCOUS (N=100)
Arrhythmia (Cardiac disorders) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 3 (3)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 (3)
Intestinal Ischaemia (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Inflammatory Marker Increased (General disorders) | 1 (1)
Multi-Organ Failure (General disorders) | 2 (2)
Stent-Graft Endoleak (General disorders) | 9 (9)
Systemic Inflammatory Response Syndrome (General disorders) | 2 (2)
Endocarditis (Infections and infestations) | 1 (1)
Graft Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1)
Vascular Bypass Dysfunction (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Compartment Syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 6 (6)
Grand Mal Convulsion (Nervous system disorders) | 1 (1)
Intracranial Aneurysm (Nervous system disorders) | 1 (1)
Neuropathy Peripheral (Nervous system disorders) | 1 (1)
Paraplegia (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Vocal Cord Paresis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aneurysm Repair (Vascular disorders) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 3 (4)
Aortic Dissection (Vascular disorders) | 3 (3)
Aortic Rupture (Vascular disorders) | 4 (4)
Arterial Thrombosis (Vascular disorders) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (3)
Haemothorax (Vascular disorders) | 1 (1)
Peripheral Artery Stenosis (Vascular disorders) | 1 (1)
Peripheral Ischaemia (Vascular disorders) | 1 (1)
Procedural Haemorrhage (Vascular disorders) | 3 (3)
Vascular Dissection (Vascular disorders) | 1 (1)
Vascular Pseudoaneurysm (Vascular disorders) | 1 (1)
Vessel Puncture Site Haematoma (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1. VCOUS (N=100)
headache (Social circumstances) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Medical Center or Investigator may, at his/her discretion, publish and/or present publicly the results of the work of Medical Center and/or Investigator performed under this Agreement. However, should Medical Center or Investigator contemplate publishing and/or presenting publicly such results, the Investigator shall provide copies of any abstracts, papers, or manuscripts to Medtronic for review at least 90 (ninety) days prior to submittal for publication or presentation.